CLINICAL TRIAL: NCT05365906
Title: Development of a Research Reference Standard for Urinary Tract Infection Using a Modified Delphi Technique
Brief Title: UTI Reference Standard: Delphi Method
Acronym: ORACLE
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Manu Bilsen, MD, MD, PhD student, Department of Infectious Diseases, Principle Investigator, Leiden University Medical Center
Other Study IDs: nWMODIV2_2022007
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Delphi-procedure consisting of four survey rounds — This study will use a modified Delphi approach, consisting of a set of iterative questionnaires. In round 1, an expert panel will grade the relevance of UTI-related items, after which a smaller core research team will compose a reference standard in a series of (online) meetings. In round 2, clinical vignettes will be used to party validate the reference standard and expert panel agreement with the new reference standard will be assessed.

SUMMARY:
This study is set up by an international core group consisting of infectious disease specialists, geriatricians, urologists, microbiologists, emergency physicians and primary care physicians to develop a consensus-based research definition of urinary tract infections. The absence of such a reference standard leads to misclassification bias and heterogeneity between studies making progress in the field of UTI difficult, for example with much needed near patient diagnostic tests.

ELIGIBILITY:
Inclusion criteria:

* Medical specialist working in the following fields: infectious diseases, urology, geriatric medicine, acute/emergency medicine, intensive care medicine, microbiology, and primary care
* Clinical and/or research experience with urinary tract infections

Exclusion criteria:

* Residency not completed yet
* Working in a different field than described above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National and international experts will be invited by email to participate in the Delphi process. Since a heterogeneous expert panel is an important feature of Delphi studies, all relevant specialties will be represented in the panel, including infectious diseases, urology, geriatric medicine, acute/emergency medicine, intensive care medicine, microbiology, and primary care. To avoid selection bias when composing the expert panel and to create a sufficiently large panel, experts will be recruited through various platforms. Experts will be allowed to invite other experts, so called 'snowballing'.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Consensus | Through study completion, an average of 7 months
  The primary study endpoint is the degree of consensus among the expert panel regarding the ORACLE reference standard.
  In round 1, consensus is defined as follows:
  An item is deemed indicative of UTI in case of a panel median of 7-9, without disagreement; uncertain in case of a panel median of 4-6 OR any median with disagreement; and not indicative of UTI in case of a panel median of 1-3, without disagreement. Disagreement exists when more than a third of responses are in the upper and the lower tertiles for the item in question
  In round 2, consensus is not predefined (i.e. with a minimum percentage). Instead, the level of agreement with a preliminary reference standard will be assessed by a dichotomous yes/no question and experts will have the possibility to give feedback on the reference standard. Thereafter, the adjusted reference standard will be presented and the level of agreement (and relative improvement) will be assessed by a dichotomous yes/no question again.

CONTACTS AND LOCATIONS:
Overall Officials: Manu Bilsen, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided